CLINICAL TRIAL: NCT00345475
Title: A Prospective Study Of Pregnancies Exposed to UCB Antiepileptic Drugs to Determine if There is a Potential Increase in the Risk of Major Birth Defects
Brief Title: UCB Antiepileptic Drugs (AED) Pregnancy Registry (Formerly the Keppra® Pregnancy Registry)
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: N01326
Record Dates: First submitted 2006-06-26; First posted 2006-06-28 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Birth Defects; Pregnancy Complications; Epilepsy; Seizures
Keywords: Birth Defects; Epilepsy; High Risk Pregnancy
MeSH Terms: conditions — Congenital Abnormalities; Pregnancy Complications; Epilepsy; Seizures

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- AED treatment: Women being treated with UCB AEDs while pregnant.

SUMMARY:
This is a prospective, observational, exposure-registration and follow-up study of women and their offspring exposed to Keppra® (levetiracetam) and Keppra XR® at the time of conception (i.e., any time from the first day of the last menstrual period) and/or during pregnancy. The UCB AED Pregnancy Registry is designed to monitor pregnancies exposed to Keppra® and Keppra XR® in order to determine if there is a potential increase in the risk of major birth defects compared to rates from women in the general US population.

The objectives of the UCB AED Pregnancy Registry are:

* To prospectively collect data concerning 1) exposure to Keppra® and Keppra XR® during pregnancy, 2) potential confounding factors, 3) outcome of pregnancy, and 4) long-term pediatric outcome
* To review reported cases of possible birth defects
* To estimate the risk of birth defects occurring in live-born offspring of women exposed to Keppra® and Keppra XR® during pregnancy

This study is being conducted in the United States (US). Enrollment in the Registry is voluntary. The UCB AED Pregnancy Registry is sponsored by UCB, Inc. and is managed by INC Research. The scientific conduct and analysis of the Registry is overseen by an Expert Panel consisting of external specialists in teratology/genetics, epidemiology, maternal and fetal medicine, and neurology (external member details available upon request).

ELIGIBILITY:
Inclusion Criteria:

The subjects must meet the following criteria for registration:

* Enroll prospectively (patient is still pregnant and no structural defects have been noted on a prenatal test)
* Exposure to Keppra® and Keppra XR® on or after the first day of the patient's last menstrual period (verified by date or gestational age of exposure)
* For patient-initiated enrollments, provide verbal or written consent to participate in the Registry
* For patient-initiated enrollments, provide contact information for herself, her HCP, and the infant's HCP (as applicable)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: See Inclusion Criteria
  - Women who have been diagnosed with Epilepsy and continued their UCB AED medication while pregnant
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2004-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The number of birth defects reported and confirmed by a teratologist | Throughout pregnancy and up to 3 years of life
  The purpose of the UCB AED Pregnancy Registry is to monitor pregnancies exposed to UCB AEDs to determine if there is a potential increase in the risk of major birth defects.

CONTACTS AND LOCATIONS:
Overall Officials: Vikki Brown, MD, Principal Investigator — Syneos Health; Jürgen Bentz, PhD, Study Director — UCB Pharma
Locations (1):
- INC Research, Wilmington, North Carolina, United States

REFERENCES:
- [Derived] Scheuerle AE, Holmes LB, Albano JD, Badalamenti V, Battino D, Covington D, Harden C, Miller D, Montouris GD, Pantaleoni C, Thorp J, Tofighy A, Tomson T, Golembesky AK. Levetiracetam Pregnancy Registry: Final results and a review of the impact of registry methodology and definitions on the prevalence of major congenital malformations. Birth Defects Res. 2019 Aug 1;111(13):872-887. doi: 10.1002/bdr2.1526. Epub 2019 May 23. PMID 31124321
- See also: Related Info — http://www.keppra.com